CLINICAL TRIAL: NCT01184183
Title: Prospective Randomized Trial Comparison of Accuseal and Bovine Pericardial Patch During Endarterectomy
Brief Title: Trial Comparison of Accuseal and Bovine Pericardial Patch During Endarterectomy
Status: Completed | Type: Observational
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Patrick Stone, MD, Patrick Stone, M.D., Vascular Center of Excellence(CAMC Medical Staff - with admitting privileges)., CAMC Health System
Other Study IDs: 09-02-2136
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Coronary Stenosis
Keywords: Patch for Carotid Endarterectomy
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Accuseal patch
  Interventions: Procedure: Comparing Accuseal Vs. Bovine Pericardial in CEA
- Bovine Pericardial patch
  Interventions: Procedure: Comparing Accuseal Vs. Bovine Pericardial in CEA

INTERVENTIONS:
Procedure: Comparing Accuseal Vs. Bovine Pericardial in CEA — Accuseal patch - The Goretex Company has since designed a new patch, "the Accuseal," which is marketed as decreasing the intra-operative time (i.e, having a short hemostasis time) without affecting the perioperative stroke rate.
  Bovine Pericardial patch - The Bovine Pericardial patch has been used for nearly two decades, since the late 1990s. However, studies based on retrospective review of data in which patients received the Bovine Pericardial patch, reported the clinical outcomes post-operative stroke, death, time to hemostasis and recurrent restenosis.

SUMMARY:
Carotid Endarterectomy (CEA), surgical removal of the blockage in the neck artery, is the accepted management of choice for significant blockage of the carotid artery. Previous studies showed improved perioperative outcomes and prevention of recurrent blockage by the use of the patch to close the surgical incision in the artery. The ideal patch reduces bleeding and prevents recurrent blockage.This is looking at long-term results toward improvement with the use Accuseal patch than Bovine Patch.

DETAILED DESCRIPTION:
This study will be a prospective, randomized, evaluation comparing the outcomes resulting from the use of two different patches (Accuseal vs Bovine Pericardial) used for CEA.Our proposed study will evaluate the perioperative (within 30 days of operation) and long-term (6 month, 1 year, 2 year, 3 year) complications associated with the Accuseal and Bovine Pericardial patches. This will include thrombosis of the carotid artery, and the degree of recurrent plaque formation of the patched artery as determined by duplex ultrasound evaluation in the perioperative and long-term periods.Patients will be blinded to the type of patch they received.Survival analysis (Kaplan-Meier) (used in this case for time to the event analysis) will be used for time to restenosis, time to stroke, and time to late death.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with >50% stenosis or Asymptomatic patients >60% stenosis: i.e.: patients experiencing a neurological event(s) such as a trans-ischemic attack, cerebrovascular accident, amaurosis fugax, and/or a preoperative duplex ultrasound, magnetic resonance angiogram, or Angiogram indicative of severe > 60% carotid artery stenosis.

Exclusion Criteria:

* will be enforced for those less than 18 years of age, patients who for religious reasons can not accept a Bovine Pericardial patch and those with a combined procedure ie: coronary artery bypass graft (CABG) and CEA.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population includes Carotid Endarterectomy (CEA), surgical removal of the blockage in the neck artery patients.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to evaluate the perioperative and long-term complications (thrombosis of the carotid artery, and the degree of restenosis of the patched artery as determined by duplex ultrasound evaluation). | within 30 days of operation,6 month, 1 year, 2 year, 3 year

SECONDARY OUTCOMES:
We hypothesize that the Accuseal patch will have a longer hemostasis time but a lower associated stroke rate and a longer time to restenosis than the Bovine Pericardial patch. | within 30 days of operation,6 month, 1 year, 2 year, 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stone, M.D., Principal Investigator — Vascular Center of Excellence(CAMC Medical Staff - with admitting privileges)
Locations (1):
- Vascular Center of Excellence, Charleston, West Virginia, United States

REFERENCES:
- [Result] Stone PA, AbuRahma AF, Mousa AY, Phang D, Hass SM, Modak A, Dearing D. Prospective randomized trial of ACUSEAL versus Vascu-Guard patching in carotid endarterectomy. Ann Vasc Surg. 2014 Aug;28(6):1530-8. doi: 10.1016/j.avsg.2014.02.017. Epub 2014 Feb 19. PMID 24561207